CLINICAL TRIAL: NCT04695002
Title: Does the Application of a Digital Tool With Real-time, Self-reported Data Facilitate Shared Decision-making and Increase Self-efficacy in Vocational Rehabilitation? A Mixed Methods Study
Brief Title: Can a Digital Tooll Facilitate Shared Decision-making and Increase Self-efficacy in Vocational Rehabilitation?
Status: Terminated | Type: Observational
Why Stopped: Too few participants enrolled due to COVID19
Sponsor: Region MidtJylland Denmark (Other)
Collaborators: Aarhus County, Denmark (Other)
Responsible Party: Principal Investigator, Nanna Rolving, Senior researcher, Region MidtJylland Denmark
Other Study IDs: A3156
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Musculoskeletal Pain
Keywords: Rehabilitation, Vocational; Telemedicine
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Citizens in the control group participate in the existing course of vocational rehabilitation offered in the municipal employment department, without the use of MIRA app.
  Interventions: Behavioral: Control
- MIRA group: Citizens in the MIRA group will participate in the existing course of vocational rehabilitation offered in the municipal department. In addition they will be introduced to MIRA at the beginning of the rehabilitation course, and use MIRA throughout the course of rehabilitation.
  Interventions: Behavioral: MIRA

INTERVENTIONS:
Behavioral: MIRA — Based on the initial assessment, the citizen and professional agree what outcomes the citizen should report in MIRA. This could be pain, mood, sleep quality, energy level, dependent on the priorities of the citizen. Similarly, different activities are reported, e.g. exercise, social activities, prolonged sitting or work-related tasks. The citizen and the professional agree how often the citizen reports the outcomes and tasks, and the citizen is notified by the MIRA-app when it's time for reporting. The data will be visualized in a graph for the professional in the back-end of the system, making it possible for the citizen and the professional to view the same, real-time reported data. This provides the base for discussing and adjusting the course of rehabilitation as symptoms change over time. At the same time, this increases the citizen's knowledge of how symptoms, mood, sleep and activities all interact, thereby giving them the tools better cope with their health condition.
  Groups: MIRA group
Behavioral: Control — Citizens in the control group participate in the standard course of vocational rehabilitation, without the use of MIRA app. Citizens are referred from the jobcenter if the case manager assesses that a health condition limits the citizen's ability to resume work. The typical course of rehabilitation lasts 4-12 weeks, and is managed by a physiotherapist, a psychologist and a physician. Depending on the condition of the citizen, the rehabilitation may be managed by only two of the three professionals. During the course of rehabilitation, the citizen may consult the team with varying frequency. If physical rehabilitation is part of the prescribed rehabilitation, the citizen shows up twice per week for several weeks of supervised exercise, whereas rehabilitation courses where self-management is in focus, only biweekly consultations may be provided. The decisions and planning of contents and duration of the rehabilitation programme is done in collaboration with the citizen.
  Groups: Control group

SUMMARY:
The study investigates both the effects and the experienced value of the mobile application, MIRA, which is a combination of an electronic diary, a dialogue tool and a decision support tool. The individual user registers real-time data reported in a mobile application, e.g. pain, sleep, mood, social activities, work-related activities, based on the goals and condition of the individual user. In this study, users are citizens participating in vocational rehabilitation due to long term sick leave.

The purpose of MIRA is to support a positive and trustful relationship between the citizen and the professional, and to enhance user involvement and shared decision making in the course of rehabilitation. This happens through promotion of the citizens knowledge and understanding of their own health condition and increase his or her self-efficacy, i.e. their ability to cope with their health condition at work and in everyday life.

The study uses a combination of quantitative and qualitative methods, analysed both individually and in combination, where findings of the different methods are combined to provide a deeper understanding of the positive and negative effects of using MIRA in vocational rehabilitation.

In this way the study investigates both the effect of applying a digital tool, such as MIRA, on a number of quantifiable measures (using questionnaires), and at the same time the study explores what works for whom and why using qualitative and combined methods. In this way, the study aims to contribute with knowledge in a balanced manner, regarding the pros and cons of using digital tools with real-time self-reported data in rehabilitation.

The study aim will be fulfilled through the following sub-purposes:

1. To investigate the effect of using MIRA in a course of vocational rehabilitation in relation to the citizens' self-efficacy for pain and work and their experience of shared decision-making in the course of rehabilitation.
2. To investigate the citizens' experience with and perception of using a digital tool like MIRA in their course of rehabilitation.
3. To investigate the professionals' experience with and perception of using a digital tool like MIRA in the course of rehabilitation.
4. To investigate the mechanisms of effect of MIRA (i.e. what works for whom and why), through and integrated analysis of the findings of sub-purpose 1-3.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a course of vocational rehabilitation at a multidisciplinary health care unit at a municipal employment department.
* On sick leave or unemployed due to musculoskeletal or stress-related disorders
* In the working age (18 - 68 years approximately)

Exclusion Criteria:

* On sick leave or unemployed for other reasons, e.g. psychiatric disorders or cancer;
* Under the age of 18 or older than 68 years (approximately)
* Not sufficiently familiar with Danish language to use the MIRA app as intended.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study takes place in a multidisciplinary health care unit in a municipal employment department in Denmark. The study population consists of citizens who referred from the job centre due to limitations in their work ability, as assessed by the case managers, due to musculoskeletal and/or stress-related disorders (the two conditions are often interrelated). In the present study only citizens with a sufficient level of Danish are included, as the MIRA-app only exists in a Danish version. Citizens are between the age of 18 and 68 (i.e, working age), and may be employed, but on prolonged sick leave, or may be unemployed.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Return-to-work Self-efficacy Scale (RTW-SE) | At baseline and at end of rehabilitation, an average of 8 weeks
  The RTW-SE is a 10-item questionnaire measuring the respondent's self-efficacy for coping with their health condition in relation to returning to work. Score ranges from 10-50 points, with 50 points reflecting the highest level of self-efficacy

SECONDARY OUTCOMES:
CollaboRATE | At end of rehabilitation, an average of 8 weeks
  CollaboRATE is a 3-item questionnaire, measuring to what extent the respondent feels involved in the decision making process in their course of rehabilitation (i.e. shared decision making) on a scale of 0-9 (worst-best). An average score of the three items is calculated
WHO-5 | At baseline and at end of rehabilitation, an average of 8 weeks
  WHO5-index is a 5-item generic questionnaire for measuring self-reported quality of life and general well-being. Each item is scored on a scale of 5 (best) to 0 (worst), adding up to a total score of 0-25

OTHER OUTCOMES:
Usability of MIRA | At the end of rehabilitation, an average of 8 weeks
  For participants in the MIRA group 4 questions regarding the usability of MIRA is applied, e.g. the need for technical support in the use of MIRA.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, PhD, Principal Investigator — Defactum, Central Denmark Region
Locations (1):
- Sociallægeinstitutionen, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
As the data are owned by the municipality participating in the study, the primary investigator/study official is not allowed to share individual participant data